CLINICAL TRIAL: NCT01067183
Title: Does a Portable Biofeedback Tool Reduce Physician Stress?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Dr Jane Lemaire, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-22185
Record Dates: First submitted 2010-02-09; First posted 2010-02-11 (Estimated); Last update posted 2010-02-19 (Estimated); Status verified 2010-02

CONDITIONS: Stress
Keywords: stress reduction; physician wellness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- breathing and biofeedback device (Experimental): This group of physicians were trained in the use of the relaxation breathing technique and the biofeedback device, and then used this portable stress reduction tool on a daily basis with twice weekly visits with the research team. After the 28 day RCT, they were invited to continue to use the device at their discretion during a trial extension from day 28-56 to see if any effect measured was maintained.
  Interventions: Behavioral: portable biofeedback tool and relaxation breathing technique
- control arm (No Intervention): This group did not undergo training in the breathing technique and use of the PSMD during the RTC trial day 0-28, but were visited twice weekly by the research team to collect outcome data. During the trial extension Day 28-56, this group did undergo a 1 hr training session with the PSMD and invited to use it at their discretion over the 28 days. Effectiveness outcome data (day 28-56) was collected at day 56.

INTERVENTIONS:
Behavioral: portable biofeedback tool and relaxation breathing technique — The intervention group were trained in relaxation breathing technique and the use of a portable biofeedback tool that informs them of the success of the technique...thus behavioral therapy using a biofeedback device
  Other Names: emwave personal stress reliever
  Arms: breathing and biofeedback device

SUMMARY:
Given the nature of their work duties and work environment, physicians often experience stress within the workplace and chronic stress negatively impacts physician wellness. Physician wellness is now linked to quality of patient care. The stress response can be broken down into four components: the stressor, the reaction, the physiological response and the experience of the physiological response. Stress can also be absolute (e.g. threat to life) and relative (e.g. I have 3 more consults to see). Stress management refers to a range of processes that are intended to mitigate one or more aspects of the psychobiology of stress. Biofeedback is a useful way of providing guidance and reinforcement for successful management of the physiological response to stress. It is important to provide physicians with effective tools for stress management. The objective of this study is to compare measures of stress and well-being among physicians allocated to learn a relaxation breathing technique and to use a biofeedback tool (referred to as a portable stress management device or PSMD) for 28 days (intervention group) and those allocated to standard care for 28 days (control group).

DETAILED DESCRIPTION:
After completion of the 28 day RCT with a control group and an intervention group, we conducted a trial extension for an additional 28 days. During that time, the original control group was trained in the use of the portable stress management device and used it, without support of the research team, for 28 days. Also during that time, the original intervention group were told that they could keep the PSMD and use it as they like. At the end of the 28 day trial extension, stress, and physiological parameters were measured again. For the initial control group, this allowed us to test effectiveness of the PSMD (real life 1 hr training on the device then unsupported use). For the initial intervention group, this allowed us to see if any effects of using the PSMD were maintained for an additional 28 days, without ongoing support from the research team.

ELIGIBILITY:
Inclusion Criteria:

* all staff physicians at the university hospital

Exclusion Criteria:

* any physician who screens positive for major depression

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Stress questionaire developed by the research team using the following resources: 1) the Sheldon Cohen Perceived Stress Scale, 2) Personal and Organizational Quality Assessment-Revised, 3) physician responses describing stress in their words. | At day 28 for RCT, at day 56 for trial extension

SECONDARY OUTCOMES:
physiological outcomes:heart rate, blood pressure, weight and salivary cortisols | At day 28 for RTC and day 56 for trial extension
physician opinions, qualitative interview data | pre and post intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Foothills Medical Center, Calgary, Alberta, Canada